CLINICAL TRIAL: NCT06787001
Title: Exploring the Interplay Between Gut Barrier and Blood-Brain Barrier Integrity, Systemic Inflammation, and Cognitive Function in Obesity
Brief Title: Understanding How Gut and Brain Barriers Are Linked to Inflammation in Obesity
Acronym: GUTBBB
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, Assoc. Prof., University Hospital, Gentofte, Copenhagen
Other Study IDs: GUTBBB
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obesity (Disorder); Systemic Inflammation Markers; Intestinal Barrier Dysfunction; Blood Brain Barrier; Neurodegenerative Disease
Keywords: intestinal barrier function; blood brain barrier function; microbiome; systemic inflammation; bacterial translocation
MeSH Terms: conditions — Obesity; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, plasma, urine, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals living with obesity: BMI > 35 kg/m2, bioimpedance-assessed body fat > 30% (men) or > 40% (women), and hip/waist-ratio > 0.85
- Individuals with lean bodies: BMI 20-25 kg/m2, bioimpedance-assessed body fat < 30% (men) or < 40% (women), and hip/waist-ratio < 0.85

SUMMARY:
The goal of this observational study is to understand how obesity affects the function of the gut and blood-brain barriers in adults. These barriers protect the body and brain from harmful substances, and changes in their function may lead to inflammation and increased risk of chronic diseases. The study will include 25 participants with obesity (BMI over 35) and 25 healthy participants (BMI 20-25) matched by age and gender.

The main questions it aims to answer are:

* How does obesity affect the blood-brain barrier and its connection to cognitive and psychopathological status?
* Does increased gut permeability lead to higher inflammation levels?
* Does obesity increase the permeability of the gut barrier?

Researchers will compare results from participants with obesity to healthy participants to determine how obesity impacts barrier function, inflammation, and overall health.

Participants will:

Attend three visits over several days, including:

* Screening visit: A health examination with weight, height, blood pressure, blood tests, and a scan to assess body fat distribution.
* Visit 1: Provide a stool sample, drink a sugar solution to assess gut permeability, collect urine samples, and take cognitive as well as psychopathological tests.
* Visit 2: Undergo an MRI scan to assess the blood-brain barrier and its function.

The study aims to identify how obesity-related changes in these barriers contribute to health risks.

DETAILED DESCRIPTION:
The study is a cross-sectional study including individuals with obesity and lean healthy controls. It is planned to recruit 25 individuals with a BMI above 35 kg/m2 and 25 lean healthy gender- and age-matched individuals with a BMI between 20-25 kg/m2. Given the extensive nature of these examinations, which include the lactulose/sucralose-mannitol test, DCE-MRI, metabolic and cognitive assessments, they will be conducted on three separate study days, in random order, and with fixed time intervals between each study day. The study employs a comprehensive approach to assess gut barrier integrity using the lactulose/sucralose-mannitol test to evaluate barrier permeability and absorptive surface area, complemented by measuring biomarkers related to gut integrity and microbial-immune interaction. Additionally, the study analyses circulating proinflammatory biomarkers and microbial genetic material to understand systemic inflammation and bacterial translocation in obesity. The integrity of the BBB is examined using DCE-MRI to detect alterations in obesity and investigate correlation between BBB permeability and obesity-related neurological conditions. Cognitive functions are assessed through tests that evaluate domains like processing speed and memory and psychopathological tests will evaluate depressive and anxiety symptoms. These tests explore the potential impact of obesity on the central nervous system. Metabolic and physiological measurements, including glucose levels, haemoglobin A1c, and body composition, provide insights into the metabolic effects of obesity and its broader physiological implications.

ELIGIBILITY:
Inclusion criteria for individuals living with obesity

* BMI > 35 kg/m2, bioimpedance-assessed body fat > 30% (men) or > 40% (women), and hip/waist-ratio > 0.85
* Age ≥40 and ≦70 years
* Sterilised or postmenopausal women (> 12 months amenorrhoea or females ≥ 60 years of age) or women who are sexually abstinent during the entire study period or are practicing non-hormonal contraception (no contraceptive pill, no hormonal intrauterine device) during the entire study period
* Able to understand written participant information and give signed informed consent.

Inclusion criteria for lean healthy controls

* BMI 20-25 kg/m2, bioimpedance-assessed body fat < 30% (men) or < 40% (women), and hip/waist-ratio < 0.85
* Age ≥40 and ≦70 years
* Sterilised or postmenopausal women (> 12 months amenorrhoea or females ≥ 60 years of age) or women who are sexually abstinent during the entire study period or are practicing non-hormonal contraception (no contraceptive pill, no hormonal intrauterine device) during the entire study period

Exclusion Criteria:

* Diagnosis of diabetes mellitus type 1 or type 2.
* Inflammatory gastrointestinal conditions such as Crohn's disease, ulcerative colitis, clinically significant food allergies, candidiasis, etc.
* Previous bariatric surgery, or surgeries involving the removal of intestinal tissue
* The use of weight loss-inducing medication such as GLP-1 receptor agonists, bupropion/naltrexone, and orlistat within 90 days prior to screening
* Planned elective surgery during the study period with the exception of dermatosurgical, ENT (ear, nose, throat) or dental procedures not requiring general anaesthesia and/or perioperative antibiotic treatment
* Chronic systemic inflammatory diseases (e.g. rheumatoid arthritis) and other conditions significantly affecting inflammation status or immunoregulation (severe allergies, status post transplantation etc.)
* History of sleep disorders
* Chronic infectious diseases such as hepatitis, HIV etc.
* Use of proton pump inhibitors, metformin, anti-biotic, lipid-lowering statins, laxatives, antihistamines, paracetamol, aspirin, statins, tricyclic antidepressants, selective serotonin reuptake inhibitor antidepressants and any other medications correlated to changes in faecal microbiome diversity for the period of the study and within 20 days prior to screening
* Active use of nicotine products, including but not limited to cigarettes, vapes, or any other form of nicotine consumption.
* Abuse of alcohol and/or drugs, or any other co-existing conditions that will make the individual unsuitable to participate in the study, as deemed by the investigators
* Pregnancy or desire to become pregnant during the study period
* Breastfeeding
* Any concomitant disease or treatment that, at the discretion of the investigators, might jeopardise the participant's safety during the study
* Mental incapacity or language barriers that preclude adequate understanding or cooperation, or unwillingness to comply with study requirements
* Body weight above the MRI scanner's maximum capacity of 140 kg or claustrophobia at a level, which makes MRI scans impossible
* Severe kidney disease with increased serum creatinine and low estimated glomerular filtration rate (GFR) (<60ml/min/1.73m2)
* Magnetic foreign objects in the body (e.g. pacemaker, metal implants from operation, etc.)
* Adherence to a restrictive diet (e.g. ketogenic diet, vegan diet, raw diet, low FODMAP diet, and paleo diet) which is significantly correlated to changes in faecal microbiome diversity 7.2.3. Criteria for discontinuation in the study
* Withdrawal of informed consent
* Pregnancy
* Any safety consideration as assessed by the investigators
* Any exclusion criterion developing or being diagnosed during the course of the study
* Non-compliance with the study protocol as deemed by the investigators

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older individuals with and without obesity
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
BBB permeability | 25 minutes post contrast administration
  Differences in BBB permeability using Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) between individuals with and without obesity

SECONDARY OUTCOMES:
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and 0-5h Lactulose/Mannitol ratio
  Ki values from DCE-MRI and Lactulose/Mannitol ratio from Lactulose/Sucralose-Mannitol test.
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and 5-24h Lactulose/Mannitol ratio
  Ki values from DCE-MRI and Lactulose/Mannitol ratio from Lactulose/Sucralose-Mannitol test.
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and baseline (fasting) Zonulin
  Ki values from DCE-MRI and quantities of plasma Zonulin
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and baseline (fasting) Citrulline
  Ki values from DCE-MRI and quantities of plasma Citrulline
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and baseline (fasting) Regenerating islet-derived protein 3-alpha
  Ki values from DCE-MRI and quantities of plasma Regenerating islet-derived protein 3-alpha
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and baseline (fasting) LBP
  Ki values from DCE-MRI and quantities of plasma Lipopolysaccharide binding protein
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and baseline (fasting) sCD14
  Ki values from DCE-MRI and quantities of plasma soluble cluster of differentiation 14
Correlation between BBB permeability and gut barrier permeability | 25 minutes post contrast administration and postprandial AUC of full blood bacterial DNA
  Ki values from DCE-MRI and full blood bacterial DNA
Correlation between BBB permeability and markers of neuronal damage | 25 minutes post contrast administration and baseline (fasting) Amyloid beta
  Ki values from DCE-MRI and quantities of plasma Amyloid beta
Correlation between BBB permeability and markers of neuronal damage | 25 minutes post contrast administration and baseline (fasting) P-Tau
  Ki values from DCE-MRI and quantities of plasma P-Tau
Correlation between BBB permeability and markers of neuronal damage | 25 minutes post contrast administration and baseline (fasting) NfL
  Ki values from DCE-MRI and quantities of plasma NfL
Correlation between BBB permeability and markers of neuronal damage | 25 minutes post contrast administration and baseline (fasting) GFAP
  Ki values from DCE-MRI and quantities of plasma GFAP
Correlation between BBB permeability and markers of neuronal damage | 25 minutes post contrast administration and baseline (fasting) Alfa-Synuclein
  Ki values from DCE-MRI and quantities of plasma Alfa-Synuclein
Correlation between BBB permeability and systemic inflammation | 25 minutes post contrast administration and baseline (fasting) HS CRP
  Ki values from DCE-MRI and quantities of plasma High sensitivity CRP
Correlation between BBB permeability and systemic inflammation | 25 minutes post contrast administration and baseline (fasting) TNF alfa
  Ki values from DCE-MRI and quantities of plasma TNF alfa
Correlation between BBB permeability and systemic inflammation | 25 minutes post contrast administration and baseline (fasting) IL 1 beta
  Ki values from DCE-MRI and quantities of plasma IL 1 beta
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and body mass index
  Ki values from DCE-MRI and Body mass index
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and bioimpedance-assessed body fat
  Ki values from DCE-MRI and bioimpedance-assessed body fat
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) Glucose
  Ki values from DCE-MRI and plasma Glucose
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) HbA1c
  Ki values from DCE-MRI and plasma HbA1c
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) Insulin
  Ki values from DCE-MRI and plasma Insulin
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) HDL cholesterol
  Ki values from DCE-MRI and plasma HDL cholesterol
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) Triglycerides
  Ki values from DCE-MRI and plasma Triglycerides
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) LDL cholesterol
  Ki values from DCE-MRI and plasma LDL cholesterol
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) VLDL cholesterol
  Ki values from DCE-MRI and plasma VLDL cholesterol
Correlation between BBB permeability and metabolic markers | 25 minutes post contrast administration and baseline (fasting) ALT
  Ki values from DCE-MRI and plasma ALT

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided